CLINICAL TRIAL: NCT03780153
Title: The Norwegian Adult Achondroplasia Study
Status: Completed | Type: Observational
Sponsor: Sunnaas Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/FO249324
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2021-12

CONDITIONS: Achondroplasia
MeSH Terms: conditions — Achondroplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Diagnosis of achondroplasia will be genetically verified. Blood samples for lipids, glucose, thyroid-, liver and kidney function and key regulating hormones in fat- and glucose metabolism
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — Observation study. No intervention

SUMMARY:
The study aims to investigate the Norwegian adult achondroplasia population regarding degree and extent of symptoms and clinical manifestations and how this population manages in daily life, including demographics, physical function, and work participation.

DETAILED DESCRIPTION:
The present study aims to investigate the degree and extent of spinal stenosis, chronic pain, sleep apnoea, impaired hearing, cardiovascular risk factors and body composition in Norwegian adults with achondroplasia. The study will also explore these factors' impact on physical function, ability to perform daily activities, work participation and needs for assistive devices and social benefits. The study is conducted in collaboration with the Norwegian Restricted Growth Association, and TRS National Resource Centre for Rare Disorders, Sunnaas Rehabilitation Hospital, Lovisenberg Hospital and Oslo University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Residents of Norway
* Aged 16 years or older
* Clinical and genetic diagnosis of achondroplasia
* Speak and understand the Norwegian language.

Exclusion Criteria:

* Severe cognitive deficits, mental illness or substance abuse
* Having a medical condition making them unable to participate in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — 16 years or older
Study Population: Adults 16 years or older with achondroplasia
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Describe the prevalence of medical complications in adults with achondroplasia | 2 years
  Describe prevalence of medical complications in a cohort of Norwegian adults with achondroplasia using interview, clinical examination and review of medical records. Data on spinal stenosis will be obtained by face-to-face interview, clinical examination, and review of medical charts including MRI-scans. Assessment of sleep apnoea will include an overnight sleep registration (polygraphy). Hearing will be assessed by standardized examination including audiometry, tympanometry and impedance measurements
Describe prevalence of cardiovascular risk factors in adults with achondroplasia, and investigate body composition. | 2 years
  Cardiovascular risk factors, including smoking habits and blood pressure, will be recorded by interview and clinical examination, and will also include a fasting blood sample for lipids, glucose, HbA1C, thyroid, kidney and liver function tests. Body composition will be assessed by anthropometric measures (height in cm, weight in kg, waist circumference in cm, and hip circumference in cm), BMI will be calculated, and body fat content and distribution will be assessed by using MRI.
Demographics and activity of daily living (ADL), education and work participation | 2 years
  Data on age, gender, education level, work participation, needs for assistive devices and social benefits will be obtained by interview. Assessment of ADL will be obtained by clinical interview and by use of The Health Assessment Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vegard Strom, Phd, Study Director — Sunnaas Rehabilitation Hospital
Locations (1):
- Sunnas Rehabilitation Hospital, Nesoddtangen, Akershus, Norway

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data will be available on request

REFERENCES:
- [Derived] Fredwall SO, Aberg B, Berdal H, Savarirayan R, Solheim J. Hearing loss in Norwegian adults with achondroplasia. Orphanet J Rare Dis. 2021 Nov 4;16(1):468. doi: 10.1186/s13023-021-02095-7. PMID 34736503
- [Derived] Fredwall SO, Overland B, Berdal H, Berg S, Weedon-Fekjaer H, Lidal IB, Savarirayan R, Manum G. Obstructive sleep apnea in Norwegian adults with achondroplasia: a population-based study. Orphanet J Rare Dis. 2021 Apr 7;16(1):156. doi: 10.1186/s13023-021-01792-7. PMID 33827611
- [Derived] Fredwall SO, Linge J, Leinhard OD, Kjonigsen L, Eggesbo HB, Weedon-Fekjaer H, Lidal IB, Manum G, Savarirayan R, Tonstad S. Cardiovascular risk factors and body composition in adults with achondroplasia. Genet Med. 2021 Apr;23(4):732-739. doi: 10.1038/s41436-020-01024-6. Epub 2020 Nov 18. PMID 33204020